CLINICAL TRIAL: NCT00382499
Title: A Prospective Evaluation of the Addition of Intraoperative Intravenous Lidocaine Infusion to General Anesthetic in Total Abdominal Hysterectomy.
Brief Title: Intraoperative Lidocaine Infusion for Analgesia (ILIA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Dr. ILIA Charapov, University of Ottawa, Departmet of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #2006512-01H
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Elective Total or Subtotal Abdominal Hysterectomy
Keywords: Intravenous Lidocaine; Lidocaine Infusion; Total Abdominal Hysterectomy; Analgesia; Anesthesia; Adjunct
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lidocaine (Experimental): IV lidocaine in OR as described in methods
  Interventions: Drug: Lidocaine Intravenous Infusion

INTERVENTIONS:
Drug: Lidocaine Intravenous Infusion — 1.5 mg/kg IV bolus on induction, 3 mg/kg/hr infusion from inducation until fascia closure

SUMMARY:
The purpose of this study is to evaluate the efficacy of intravenous lidocaine infusion administered during general anesthesia in:

1. Reducing length of hospital stay following total abdominal hysterectomy
2. Reducing postoperative analgesic requirement following total abdominal hysterectomy.

Hypothesis:

The addition of an intraoperative lidocaine infusion to a balanced anesthetic technique will result in up to 50% of patients being discharged after postoperative day 2 compared with the current 21%. Also, it will result in a 30% reduction in opiod consumption during the first 48 hours following total abdominal hysterectomy.

Assumption:

Patients in the intervention and control groups will be titrated to approximately equal analgesia because they will self-administer enough pain-controlling medications to make their postoperative pain experience the same.

Primary outcomes:

1. Length of hospital stay
2. Total opioid use at 48 hours postoperatively

Secondary outcomes. The following data will be collected and analyzed:

1. Intraoperative data: BIS scores (to control depth of anesthesia); intraoperative serum lidocaine levels; intraoperative opioid use
2. Opioid use in the recovery room
3. Patient Controlled Analgesia (PCA) morphine requirements postoperatively up to 48 hours
4. Oral pain controlling medication use up to 48 hours postoperatively if IV PCA discontinued before 48 hours
5. Verbal Analogue Scale (VAS) pain scores in recovery room and during first 2 days post-operatively
6. Incidence of side effects that can be attributed to local anesthetic toxicity
7. Incidence of nausea and vomiting and anti-emetic use up to 48 hours postoperatively
8. Time of first flatus and first bowel movement.

DETAILED DESCRIPTION:
Provide the rationale for the study (see list of references attached separately).

Provide the rationale for the study (see list of references attached separately).

Adequate postoperative pain control is still a major problem for many surgical patients. Identifying better ways of controlling pain during and after surgery remains an ongoing goal of research in anesthesia. Continuous infusion of IV lidocaine has been identified in the anesthetic literature as a valuable supplement to general anesthesia. Approximately 20% of all total abdominal hysterectomies at The Ottawa Hospital today are done using a continuous IV lidocaine infusion in addition to general anesthesia. Considering its low cost, ease of administration, and low incidence of side effects, lidocaine presents an attractive anesthetic option.

However, there have been only a few randomized controlled trials to date that have assessed the effect of IV lidocaine on a patient's pain control. These trials were small single center studies that require independent validation at other institutions and in other surgical populations. In the previous trials, the standard anesthetic technique was not as well controlled as it will be in this trial. If approved this study will add to the scant but promising literature concerning peri-operative lidocaine use for analgesia.

1. Lidocaine infusion supplements general anesthesia and improves analgesia. Lidocaine has been used to supplement general anesthesia for over 50 years (1). It has a MAC sparing effect that allows reduction of other anesthetic agents in a balanced anesthetic technique (1). Lidocaine infusions improve pain scores in burn patients and provide sufficient analgesia without the addition of an opioid analgesic (3). Its use is well established in chronic neuropathic and ischemic pain (6,7). Over the last decade, its use in the management of acute pain and pre-emptive analgesia has increased. Studies demonstrating improved pain scores with movement and at rest in major abdominal surgeries and radical retropubic prostatectomy have been published (2,5,8).
2. IV Lidocaine infusion dose and toxicity (2,3,4,5,6,7,10). Lidocaine toxicity does not occur with plasma levels below 5 mcg/mL. Currently reported dosing vary between 'no IV bolus' to 3 mg/kg/hr IV bolus followed by 1.5 to 3 mg/kg/hr infusion rates. These doses generally result in plasma levels of 1.3-3.7 mcg/mL. There is no increase in local anesthetic toxicity at these plasma levels compared to placebo. In one study up to 2.6 mg/kg/hr of lidocaine had been infusing for 24 hours after the end of surgery with no reported side effects attributed to local anesthetic toxicity (4).

   In another lidocaine dose-response study an infusion of 500 mg of lidocaine over one hour in 13 patients with neuropathic chronic pain (6) resulted in plasma levels of 2.43 +/- 1.01 mcg/mL at the initial onset of analgesia. This corresponds to infusion rates of approximately 6-7 mg/kg/hr of lidocaine (no bolus). The amount of lidocaine used at the onset of analgesia was 123+/-55 mg over ~ 9-20 minutes. Complete analgesia was reported in 10 out 13 patients with corresponding plasma levels of 3.79+/- 1.00 mcg/mL with a total lidocaine dose of ~ 375 +/- 23mg over 36-54 minutes. In 3 patients there was a significant reduction in pain but no complete analgesia. Light-headedness at some time during infusion was reported in 6 out of 13 patients and their lidocaine levels ranged from 0.9 to 3.08 mcg/mL. At no time did the infusion need to be adjusted because of subjective complaints of toxicity.

   The dose of lidocaine currently used at the Ottawa Hospital Department of Anesthesia to supplement general anesthesia is a bolus of 1-1.5 mg/kg followed by an intraoperative infusion of 1.2 to 3 mg/kg/hr. In this study we propose a bolus of 1.5 mg/kg followed by 3 mg/kg/hr infusion.
3. Lidocaine infusion reduces opiod consumption. Lidocaine infusions have decreased the opioid and NSAID use following major surgery (2,5). A protocol and a case report in burn patients demonstrate markedly reduced requirements for opioid analgesia (3). The reduced use of opiods should be associated with lower incidence of opiod-related side effects and decreased use of medication to treat these side effects.
4. Lidocaine infusion improves bowel function. Lidocaine use speeds the return of bowel function that is a major complication of intra-abdominal operations. In both radical prostatectomy and cholecystectomy patients' time to passage of first postoperative bowel movement was decreased (4,5).
5. Lidocaine infusion leads to quicker discharge. Lidocaine use led to faster discharge from hospital in-patients undergoing radical prostatectomy (5). This result is likely due to the combined beneficial effects as outlined above.

Protocol:

Patients will be recruited through multiple mechanisms. These will include, but not be restricted to: preoperative assessment clinics, physicians' clinics, and hospital wards.

Anesthesia physicians, Obstetrics and Gynecology physicians, residents, and nurses involved in the care of potential total abdominal hysterectomy (TAH) candidates will be be informed about the study by primary investigators through memos, presentatations, departmental meetings. Potential subjects will be identified by these physicians, residents, and nurses involved in the care of TAH patients. Study personnel will be contacted to determine patient eligibility for the study.

Primary investigators at the Civic and General campuses of Ottawa Hospital and physicians at the Preoperative Assessment Unit (PAU) at both campuses will identify patients undergoing elective total abdominal hysterectomy. These patients will be offered an opportunity to participate in the study during standard pre-anesthetic assessment at the Pre-Admission Unit by an anesthesiologist. During this assessment a full medical history, a complete physical exam, and appropriate investigations will be carried out.

If a patient is willing to consider participation, a study investigator or their delegate will discuss the study. The study information sheet will be provided to the patient. The rationale for the study and the study protocol would be discussed using the language appropriate for the patient's background. A discussion of benefits and risks associated with the study and possible anesthetic techniques will be carried out and all questions answered at this time.

Patient consent. Once identified and their eligibility confirmed patients will be asked to provide informed written consent using the Information sheet and Consent form (Appendix 1). Participation will be entirely voluntary. Patients will neither be coerced nor offered incentives to participate.

If the patient decides to participate a Study Checklist will be completed by research personnel and placed on patient's chart. The Study Checklist form will contain pre-calculated doses of medications for that particular patient as well as concise protocol checklist for the attending anesthetist.

Randomization. Patients will be randomized using a computer generated random number table. All patients randomized will be followed and analyzed in the group to which they are allocated. All patients will be randomized as close to the time of surgery as possible to avoid randomizing patients who subsequently have surgery postponed or cancelled.

Allocation concealment: Allocation to intervention or control groups will be printed on cards placed in sealed, opaque, sequentially-numbered envelopes. Trial envelopes will be kept with research personnel and opened in numerical order when the patient has met the eligibility criteria and is ready to be randomized. An anesthesia resident or staff not involved with care of the patient will open an envelope for that patient and prepare four syringes:

* One 10mL Study Drug Bolus syringe containing either Normal Saline or 2% Lidocaine;
* Three 20mL Study Drug Infusion syringes containing either Normal Saline or 2% lidocaine.

Maintenance of confidentiality. All records will be kept confidential. Records will be kept in a locked cabinet in the Department of Anesthesiology, Civic Campus for fifteen (15) years following enrollment of the last patient. Access will be restricted to study investigators and research assistants. Data will be stored on a secure, password-protected computer within the Department of Anesthesiology and kept strictly confidential. No information capable of identifying a study participant will appear in study reports or publications

Study design: This is a prospective, randomized, double blinded, clinical trial comparing intravenous lidocaine infusion plus general anesthesia with general anesthesia alone. The intervention group will receive a balanced anesthetic with the addition of lidocaine as outlined in the anesthetic protocol outlined in appendix 2. The control group will receive a balanced anesthetic with the addition of normal saline as outlined in the appendix 2. The patients, clinicians, and study personnel will be blinded to group allocation.

Primary objectives:

1. To study the effect of the addition of intraoperative intravenous lidocaine infusion (1.5 mg/kg IV bolus followed by 3 mg/kg/hr infusion) to a balanced general anesthetic on length of hospital stay after total abdominal hysterectomy;
2. To study the effect of the addition of intraoperative intravenous lidocaine infusion (1.5 mg/kg IV bolus followed by 3 mg/kg/hr infusion) to balanced general anesthetic on opioid requirements intraoperatively, in the recovery room, and up to 48 hours post operatively.

Secondary objectives:

1. Post-operative visual analogue scale (VAS) pain scores for 48 hours;
2. Incidence of opioid related side effects including: (a) post-operative nausea and vomiting (b) subsequent anti-emetic medication use (c) decreasing time to first flatus and bowel movement;
3. Following data will also be analyzed:

   * Intraoperative lidocaine levels;
   * Incidence of side effects that can be attributed to local anesthetic toxicity;
   * Oral pain medications use up to 48 hours postoperatively if IV PCA discontinued before 48 hours.

Baseline Assessment: All patients eligible for the trial will have the following information documented preoperatively: age, sex, height, weight, body mass index, serum creatinine, calculated creatinine clearance (Cockroft-Gault), primary diagnosis, and scheduled procedure.

Management of anesthesia: All patients will undergo a standardized anesthetic according to the Study Checklist (Appendix 2) that will be completed as soon as the patient is enrolled in the study. The Study Checklist will accompany the anesthetic record and the patient to the OR. This Study Checklist will form the basis for the dosing of all the medications for the anesthetic and the order the protocol is to be completed in. The drugs that are variable in their dosing will include: propofol (will be given to the desired effect at anesthesia induction); rocuronium (will be given to the desired effect of muscle relaxation); and desflurane (will be titrated to a BIS reading of 40 to ensure adequate anesthetic depth). If needed, morphine will be available to the attending anesthesiologist should the patient demonstrate clinical signs of inadequate analgesia during the anesthetic.

Management of intervention group: Patients in the intervention group will receive lidocaine 1.5 mg/kg as part of their induction. The lidocaine bolus will be followed be a continuous intravenous infusion at 3.0 mg/kg/hr. The rate is pre-calculated and appears on the Study Checklist (Appendix 2). The infusion of lidocaine and fentanyl will be stopped upon skin closure.

Serum lidocaine levels will be collected at two points of the study:

* 30 minutes after the initial bolus
* and during surgical closure, just prior to stopping the infusion.

Management of control group: Patients in the control group will receive normal saline as part of their induction. The normal saline bolus will be followed be a continuous intravenous infusion. The rate is pre-calculated and appears on the Study Checklist (Appendix 2). The infusion of normal saline and fentanyl will be stopped upon skin closure.

Serum lidocaine levels will be collected at two points of study:

* 30 minutes after the initial bolus
* and during surgical closure, just prior to stopping the infusion.

Management of inadequate analgesia: Patients in the post anesthesia care unit (PACU) will be given their patient controlled analgesia (PCA) after immediate assessment of visual analogue scale (VAS) pain scores are complete. They can self administer morphine until their desired comfort level is reached with the help of the nurse if needed.

Management of opioid related side effects: Patients with satisfactory analgesia but experiencing unwanted sedation will be assessed by a study physician. Patients experiencing hypotension, will be given a 500mL crystalloid bolus and will assessed by a study physician. Patients with significant respiratory depression will be given naloxone in 40μg boluses until respiratory rate is >10 and will be sedation will assessed by a study physician. Patients experiencing pruritis, nausea, or insomnia will be managed with the medications outlined in the Study Checklist (Appendix 2) and these orders will be on the APS order sheet that will have been completed with the Study Checklist at the time of enrollment.

Postop care: Patients will be discharged to the ward with care as per current Total Abdominal Hysterectomy (TAH) care map.

Description of Tests: In addition to the usual bloodwork involved during this type of procedure, the anesthesiologist will collect 2 blood samples to test the levels of lidocaine in your blood during surgery. There will be no further tests.

Switching to oral analgesia: Patients who are nearing discharge criteria and being able to tolerate medications PO will be offered discontinuation of IV PCA and a switch to PO morphine 5-10 mg PO PRN q 2 hours. Patients will continue receiving Celebrex 200 PO q12hr with food intake and Tylenol 650mg PO q4hr while awake until 72 hours postop.

Discharge criteria: Patients will be discharged according as per the current discharge criteria for the care map of TAH patient at The Ottawa Hospital.

1. Adequate pain control
2. Vital signs stable
3. Afebrile (no fever)
4. Passing flatus (passing gas)
5. No or scant vaginal discharge
6. Incision clean, dry, intact, and edges approximated
7. Tolerates diet as ordered
8. Understands: staple removal instructions if applicable; New medications; discharge instructions per patient information booklet; follow-up plan with Gynecology physician
9. Understands there will be a follow up phone call in about one week by one of study investigators to assess level of satisfaction

The Gynecology physicians will make assessment for discharge eligibility daily in the first half of the day. Should the patient discharge be delayed due to logistical reasons (e.g. was ready for discharge on POD2, but seen late on POD2 and discharged home POD3) - a note of that will be made by study nurse in the study data sheet for that patient.

Post discharge follow-up: patients will be contacted by study coordinator or study nurse in approximately one week by phone to evaluate patient satisfaction with the overall experience.

Outcome assessment:

Primary outcome measure: The length of hospital stay in days will be recorded. The morphine consumption will be recorded from the PCA pump database on departure from the PACU and every 8 hours until 48 hours postoperatively. Any other opioid medication used for weaning off PCA will also be recorded and converted to morphine equivalents for analysis during the first 48 hours. This data will be compared between the two groups.

Secondary outcome measures: Post-operative visual analogue scale (VAS) pain scores will be recorded on departure from the PACU and every 8 hours until 48 hours postoperatively. The incidence of opioid related side effects will be recorded. This will include post-operative nausea and vomiting, subsequent anti-emetic medication use, time to first flatus and bowel movement. This data will be compared between the two groups.

Lidocaine levels that were measured at 30 minutes intraoperatively and just prior to the end of the infusion will also be collected and reported.

Data analysis: The number of patients discharged on post-operative day 2 will be analyzed with a chi-square analysis. The morphine consumption at 24 and 48 hours, will be analyzed with the unpaired student's t-test. Post-operative visual analogue scale (VAS) pain scores will be analyzed for statistical difference using an unpaired student's t-test. Analyses of secondary outcomes such as immediate post-operative nausea and vomiting, subsequent anti-emetic usage, time to first bowel movement will be analyzed with the unpaired student's t-test Statistical significance will be assigned a probability of <0.05 for all analyses.

Data management. Data will be recorded on standardized data collection forms. Data will be transferred from the forms to an Excel 2002 spreadsheet (Microsoft Corp, Redmond WA) at which time patients will be assigned and identified by a unique trial number. Data will be exported to SPSS 11.0.1 (SPSS Inc, Chicago Il) for analysis.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective total abdominal hysterectomy at The Ottawa Hospital and able to give informed consent.

Plus:

1. Age 30-69 inclusive;
2. ASA (American Society of Anesthesiologists) class I or II patient: (I - healthy with no systemic disease, II - systemic disease with no functional limitation);
3. Body Mass Index (BMI) of 18.5-30.

Exclusion Criteria:

Patients undergoing elective total abdominal hysterectomy at The Ottawa Hospital and unable to give informed consent., unable to provide informed consent, or unable to use patient controlled analgesia.

Plus:

1. Patients under age 30 or over age 70;
2. ASA III, IV and V class patients (III - systemic disease causing functional impairment; IV - systemic disease that is a constant threat to life; V - not expected to survive with or without surgery);
3. Obese patients (BMI>30) or undernourished (BMI<18.5) (9);
4. Unable to use patient controlled analgesia;
5. Any history of liver dysfunction;
6. Renal insufficiency defined as a creatinine clearance <50mL/min as calculated using the Cockroft-Gault formula (11);
7. History of seizure disorder;
8. Hypersensitivity or allergy to amide type local anesthetics;
9. Hypersensitivity or allergy to any of the following opiods: morphine, hydromorphone, meperidine, fentanyl;
10. Any chronic pain syndromes or opioid use greater than once per week.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay
Total opioid use at 48 hours postoperatively

SECONDARY OUTCOMES:
Intraoperative data: BIS scores (to control depth of anesthesia)
Intraoperative serum lidocaine levels
Intraoperative opioid use
Opioid use in the recovery room
Patient Controlled Analgesia (PCA) morphine requirements postoperatively up to 48 hours;
Oral pain controlling medication use up to 48 hours postoperatively if IV PCA discontinued before 48 hours;
Verbal Analogue Scale (VAS) pain scores in recovery room and during first 2 days post-operatively;
Incidence of side effects that can be attributed to local anesthetic toxicity;
Incidence of nausea and vomiting and anti-emetic use up to 48 hours postoperatively;
Time of first flatus and first bowel movement.

CONTACTS AND LOCATIONS:
Overall Officials: ILIA Charapov, MD, Principal Investigator — The Ottawa Hospital, Dept of Anesthesia; Greg Bryson, MD, Study Chair — The Ottawa Hospital, Dept of Anesthesia
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Bryson GL, Charapov I, Krolczyk G, Taljaard M, Reid D. Intravenous lidocaine does not reduce length of hospital stay following abdominal hysterectomy. Can J Anaesth. 2010 Aug;57(8):759-66. doi: 10.1007/s12630-010-9332-2. Epub 2010 Jun 8. PMID 20532723